CLINICAL TRIAL: NCT06372119
Title: Letrozole-stimulated Cycle Strategy Versus Artificial Cycle Strategy for Endometrial Preparation in Women With Irregular Menstrual Cycles: A Randomized Controlled Trial
Brief Title: Letrozole-stimulated Cycle Strategy Versus Artificial Cycle Strategy (LETSACT)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mỹ Đức Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13/23/DD-BVMD
Record Dates: First submitted 2023-12-27; First posted 2024-04-17 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Embryo Transfer; Irregular Menstruation; Letrozole; Hormone Replacement Therapy
Keywords: Blastocyst Transfer; Irregular Menstruation; Letrozole; Hormone Replacement Therapy
MeSH Terms: conditions — Menstruation Disturbances | interventions — enkephalinamide-Leu, Tyr sulfate(1)-

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Letrozole-stimulated cycle strategy (LETS) (Active Comparator): to fourth day of the menstrual cycle.
  Post-letrozole, ultrasound checks follicle growth. If ≥18mm, Ovitrelle® 250 mcg (Merck, Kenilworth, New Jersey, USA) induces ovulation.
  Luteal phase support with vaginal micronized progesterone (Cyclogest® 400 milligrams, Actavis, UK or Utrogestan® 200 milligrams, Besins, Belgium) 800 milligrams/day starting two days post-hCG.
  Embryo transfer, 5 days post-progesterone. Ultrasounds use Samsung HS-30, vaginal probe, and ≥7.5MHz frequency. Hormonal support until the 12th gestational week with vaginal micronized progesterone 800 milligrams/day.
  Cycle cancellation criteria: no follicle development on day 21 from the day of starting letrozole, spontaneous ovulation, letrozole intolerance, fluid retention. Cycle cancellation will be noted as a study's outcome.
  Interventions: Procedure: Letrozole-stimulated cycle strategy
- Artificial cycle strategy (AC) (Active Comparator): Oral estradiol valerate (Progynova® 2 milligrams, Bayer Pharma AG, Germany or Valiera® 2 milligrams, Laboratories Recalcine, Chile) 6 milligrams/day for 10 days, starting on the second to fourth day of the menstrual cycle.
  Post-estradiol, ultrasound checks endometrial thickness. If ≥7mm, start vaginal micronized progesterone (Cyclogest® 400 milligrams, Actavis, UK or Utrogestan® 200 milligrams, Besins, Belgium) 800 milligrams/day. If <7mm, increase the dose of oral estradiol valerate to 8 milligrams/day (5-6 days) and 12 milligrams/day (5-6 days).
  Embryo transfer, 5 days post-progesterone. Ultrasounds use Samsung HS-30, vaginal probe, and ≥7.5MHz frequency. Hormonal support until the 12th gestational week with vaginal micronized progesterone 800 milligrams/day.
  Cycle cancellation criteria: endometrial thickness <7mm on day 21 of using estradiol, spontaneous ovulation, oral estradiol valerate intolerance, fluid retention. Cycle cancellation will be noted as a study's outcome.
  Interventions: Procedure: Artificial cycle strategy

INTERVENTIONS:
Procedure: Letrozole-stimulated cycle strategy — Letrozole (Femara® 2.5 milligrams, Novartis, Switzerland or Lezra® 2.5 milligrams, Actavis, Rumani) 5 milligrams/day for 5 days, starting on the second to fourth day of the menstrual cycle.
  Post-letrozole, ultrasound checks follicle growth. If ≥18mm, Ovitrelle® 250 mcg (Merck, Kenilworth, New Jersey, USA) induces ovulation.
  Luteal phase support with vaginal micronized progesterone (Cyclogest® 400 milligrams, Actavis, UK or Utrogestan® 200 milligrams, Besins, Belgium) 800 milligrams/day starting two days post-hCG.
  Embryo transfer, 5 days post-progesterone. Ultrasounds use Samsung HS-30, vaginal probe, and ≥7.5MHz frequency. Hormonal support until the 12th gestational week with vaginal micronized progesterone 800 milligrams/day.
  Cycle cancellation criteria: no follicle development on day 21 from the day of starting letrozole, spontaneous ovulation, letrozole intolerance, fluid retention. Cycle cancellation will be noted as a study's outcome.
  Other Names: LETS
  Arms: Letrozole-stimulated cycle strategy (LETS)
Procedure: Artificial cycle strategy — Oral estradiol valerate (Progynova® 2 milligrams, Bayer Pharma AG, Germany or Valiera® 2 milligrams, Laboratories Recalcine, Chile) 6 milligrams/day for 10 days, starting on the second to fourth day of the menstrual cycle.
  Post-estradiol, ultrasound checks endometrial thickness. If ≥7mm, start vaginal micronized progesterone (Cyclogest® 400 milligrams, Actavis, UK or Utrogestan® 200 milligrams, Besins, Belgium) 800 milligrams/day. If <7mm, increase the dose of oral estradiol valerate to 8 milligrams/day (5-6 days) and 12 milligrams/day (5-6 days).
  Embryo transfer, 5 days post-progesterone. Ultrasounds use Samsung HS-30, vaginal probe, and ≥7.5MHz frequency. Hormonal support until the 12th gestational week with vaginal micronized progesterone 800 milligrams/day.
  Cycle cancellation criteria: endometrial thickness <7mm on day 21 of using estradiol, spontaneous ovulation, oral estradiol valerate intolerance, fluid retention. Cycle cancellation will be noted as a study's outcome.
  Other Names: AC
  Arms: Artificial cycle strategy (AC)

SUMMARY:
The goal of this randomized clinical trial is to evaluate the effectiveness of the letrozole-stimulated cycle strategy versus the artificial cycle strategy for endometrial preparation in women with irregular menstrual cycles after one cycle of endometrial preparation. The primary question it aims to answer is:

• Does the letrozole-stimulated cycle strategy for endometrial preparation result in a higher live birth rate compared to the artificial cycle strategy in women with irregular menstrual cycles after one cycle of endometrial preparation?

Participants will undergo screening before endometrial preparation for frozen embryo transfer, following which they will be randomly assigned to one of two groups: LETS or AC. In the LETS group, investigators will prescribe letrozole 5 milligrams/day for 5 days to stimulate follicular development and micronized progesterone 800 milligrams/day for luteal phase support. In contrast, the AC group will receive oral estradiol valerate 6-12 milligrams/day and micronized progesterone 800 milligrams/day. Researchers will compare the LETS and AC groups to determine if there are differences in live birth rates.

DETAILED DESCRIPTION:
Freeze-all and later frozen embryo transfer (FET) to reduce the risk of ovarian hyperstimulation syndrome (OHSS) is a common strategy in modern assisted reproduction technology (ART). Preparing the endometrium for FET in women with irregular menstrual cycles poses a challenge due to limited protocol options. There are two basic endometrial preparation regimens before FET: artificial cycle (AC) or natural cycle (NC). NC is often only considered if the woman has regular ovulation. In women with irregular menstrual cycles, the most popular conventional technique of endometrial preparation is AC. The advantages of AC include its convenience (meaning that the window of implantation can be determined actively and correctly) and its adaptability (meaning that the duration and the dose of exposure to estradiol and progesterone hormones can be flexibly scheduled). On the other hand, artificial exogenous estradiol levels may diminish endometrial receptivity, increase the risk of thrombosis and cancer, and negatively impact the baby's outcomes. Furthermore, the absence of the corpus luteum and its products in early pregnancy may be associated with an increased risk of placentation deficiency and an increased risk of (pre)eclampsia, which is already common in this population.

The current modern approach in endometrial preparation is to create the endometrial proliferative phase that mimics the NC's physiology and to attempt to produce the corpus luteum. Previous studies showed that in the general population, ovulation-based cycles resulted in considerably greater pregnancy rates than AC, regardless of whether ovulation was natural or inducted. Exogenous gonadotropins, clomiphene citrate (CC), and aromatase inhibitors (AI) are the three types of ovulation-inducing agents widely utilized for women with irregular menstrual periods. Gonadotropin is not patient-friendly due to the route of administration and increases the risk of OHSS. CC is well-known for its antagonistic effect on estrogen receptors and its negative impact on endometrial receptivity. Letrozole, a preferred drug in the AI group, has been explored for almost two decades to avoid the drawbacks of other methods. First, letrozole can stimulate mono-follicular growth and minimize the incidence of OHSS at a low cost and in a more patient-friendly manner. Second, letrozole decreases intraovarian and serum estrogen levels, thereby upregulating endometrial estrogen receptors, increasing endometrial sensitivity to estrogen increase, and preventing premature progesterone action, which results in increased endometrial proliferation. Thirdly, there was evidence that letrozole may improve endometrial receptivity by modulating the formation of αvβ3 and HOXA10 integrin, leukemia inhibitory factor (LIF), L-selectin, and pinopode formation.

The findings of some previous studies showed that the letrozole-stimulated cycle was superior to AC in terms of improving clinical pregnancy rate, live birth rate, and lower risk of miscarriage, preterm birth, pre-ecclampisa and also decreasing the risk of ectopic pregnancy. However, there was also evidence that shows no consistent advantage of letrozole as compared to AC. Notably, prior research on the effectiveness of letrozole in endometrial preparation for FET was predominantly retrospective. There were few randomized controlled trials (RCT) comparing the letrozole-stimulated cycle versus AC. However, these studies found similar treatment outcomes with two endometrial preparation methods. The sample size was also limited (N < 150), and letrozole was often used in combination with hMG concurrently.

This study will be undertaken at IVFMD, a reproductive center of My Duc Hospital in Ho Chi Minh City, Vietnam, to provide evidence on how effective letrozole is compared to conventional AC.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 - 42.
* Irregular menstrual cycle (< 21 days or > 35 days or < 8 cycles/years).
* Indicated for endometrial preparation.
* Transfer of only one blastocyst.
* Not participating in any other trials.

Exclusion Criteria:

* Allergy to letrozole or Ovitrelle or oral estradiol valerate or micronized progesterone
* Having embryos from either oocyte donation or PGT (pre-implantation genetics testings) cycles.
* Ovarian cysts that are unrelated to the oocyte pick-up.
* Confirmed diagnosis with recurrent pregnancy loss (RPL) according to ESHRE guideline 2023, recurrent implantation failure (RIF) according to ESHRE 2023 good practice recommendations.
* Endometrial abnormalities include endometrial hyperplasia, intrauterine adhesions, endometrial polyp, and chronic endometritis.
* Uterine abnormalities include leiomyomas L0, L1, or L2 (according to FIGO 2011); adenomyosis (according to MUSA 2022); congenital uterine abnormalities, include didelphus, arcuate, unicornuate, bicornuate, septate (according to ASRM 2021).
* Untreated hydrosalpinx.

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 790 (Estimated)
Dates: Start 2024-04-22 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Live birth rate after one cycle of endometrial preparation | After 22 completed weeks of gestational age.
  Live birth will be defined as the complete expulsion or extraction from a woman of a product of fertilization, after 22 completed weeks of gestational age; which, after such separation, breathes or shows any other evidence of life, such as heart beat, umbilical cord pulsation or definite movement of voluntary muscles, irrespective of whether the umbilical cord has been cut or the placenta is atached. A birth weight of 500 grams or more can be used if gestational age is unknown. Twin and higher multiple births will be reported as a single live birth event.

SECONDARY OUTCOMES:
Positive pregnancy test after one cycle of endometrial preparation | At 11 days after blastocyst transfer.
  Defined as serum human chorionic gonadotropin level greater than 25 mIU/mL.
Clinical pregnancy after one cycle of endometrial preparation | First ultrasound before 6 weeks of gestational age.
  Diagnosed by ultrasonographic visualization of one or more gestational sacs or definitive clinical signs of pregnancy at 6 weeks or more after the onset of last menstrual period. In addition to intra-uterine pregnancy, it includes a clinically documented ectopic pregnancy.
Ongoing pregnancy after one cycle of endometrial preparation | After 12 weeks of gestational age.
  Defined as pregnancy with a detectable heart rate at 12 weeks gestation or beyond.
Multiple pregnancy after one cycle of endometrial preparation | Ultrasound at 6-9 weeks of gestational age.
  Defined as the presence of more than one gestational sac at early pregnancy ultrasound (6-9 weeks gestation) (Hecher and Diehl, 2009).
Implantation rate after one cycle of endometrial preparation | Ultrasound at 6-9 weeks of gestational age.
  A cycle in which monitoring has been initiated with the intention to treat but which did not proceed to embryo transfer (as defined above).
Cycle cancellation rate | During the intervention (on day 21 from the day of starting to use letrozole or valiera).
  A cycle in which monitoring has been initiated with the intention to treat but which did not proceed to embryo transfer due to the criteria defined above or protocol violation.
Ectopic pregnancy rate after one cycle of endometrial preparation | Ultrasound at 6-9 weeks of gestational age.
  A pregnancy outside the uterine cavity, diagnosed by ultrasound, surgical visualization or histopathology.
Threatened miscarriage rate before 12 weeks of gestation after one cycle of endometrial preparation | At 12 weeks of gestational age.
  Vaginal bleeding before 12 weeks of gestation.
Early miscarriage rate after one cycle of endometrial preparation | At 12 weeks of gestational age.
  Spontaneous loss of pregnancy up to 12 weeks of gestation (Oxford Textbook of Obstetrics and Gynaecology, 2020).
Late miscarriage rate after one cycle of endometrial preparation | At 22 weeks of gestational age.
  Spontaneous loss of pregnancy between12 to 22 weeks of gestation (Oxford Textbook of Obstetrics and Gynaecology, 2020).
Gestational age at birth | On the day of delivery.
  Calculated by gestational age of all live births
Onset of labor | On the day of delivery.
  Spontaneous, labor induction, elective C-section.
Mode of delivery | On the day of delivery.
  Vaginal delivery, C-section (elective, suspected fetal distress, non-progressive labor).
Very low birth weight | On the day of delivery.
  Birth weight less than 1500g.
Low birth weight | On the day of delivery.
  Birth weight less than 2500g.
High birth weight (macrosomia) | On the day of delivery.
  Implies growth beyond an absolute birth weight, historically 4000 g or 4500 g, regardless of the gestational age ("Macrosomia: ACOG Practice Bulletin, Number 216," 2020).
Very high birth weight (macrosomia) | On the day of delivery.
  Birth weight over than 4500 g for women with diabetes, and a threshold of 5000 g for women without diabetes ("Macrosomia: ACOG Practice Bulletin, Number 216," 2020).
Gestational diabetes (GDM) | At 24-28 weeks of gestational age.
  Diagnosed according to the latest version of ADA guidelines: a 75-g OGTT, with plasma glucose measurement when patient is fasting and at 1 and 2 h, at 24-28 weeks of gestation in women not previously diagnosed with diabetes; fasting: 92 mg/dL (5.1 mmol/L); 1h: 180 mg/dL (10.0 mmol/L); 2h: 153 mg/dL (8.5 mmol/L).
Hypertensive disorders of pregnancy | On the day of delivery.
  Comprising pregnancy-induced hypertension (PIH), pre-eclampsia/eclampsia and Hemolysis, elevated liver enzymes, and low platelet count (HELLP) syndrome. PIH diagnosed after 20 weeks' gestation; systolic blood pressure ≥140 mmHg or diastolic pressure ≥90 mmHg on two occasions, two hours apart, or severely elevated single blood pressure measurement requiring an hypertensive medication. Pre-eclampsia/eclampsia diagnosed according to ACOG practice bulletin (ACOG Committee on Obstetric Practice, 2002). Diagnosis and management of preeclampsia and eclampsia. HELLP syndrome is defined as a condition with the clinical presentation of hemolysis, elevated liver enzymes, and low platelet count; lactate dehydrogenase (LDH) elevated to 600 IU/L or more, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) elevated more than twice the upper limit of normal, and the platelets count less than 100000 × 10^9/L (ACOG Committee on Obstetric Practice, 2002).
Preterm birth | On the day of delivery.
  Defined as delivery at <24, <28, <32, <37 completed weeks. A birth that takes place after 22 weeks and before 37 completed weeks of gestational age.
Stillbirth | On the day of delivery.
  The death of a fetus prior to the complete expulsion or extraction from its mother after 28 completed weeks of gestational age. The death will be determined by the fact that, after such separation, the fetus does not breathe or show any other evidence of life, such as heartbeat, umbilical cord pulsation, or definite movement of voluntary muscles. Note: It includes deaths occurring during labor.
Antepartum hemorrhage | On the day of delivery.
  Defined as bleeding from or into the genital tract, occurring from 24 weeks of pregnancy and prior to the birth of the baby (Royal College of Obstetricians and Gynaecologists, 2011).
Postpartum hemorrhage | On the day of delivery.
  Defines as cumulative blood loss greater than or equal to 1,000 mL or blood loss accompanied by signs or symptoms of hypovolemia within 24 hours after the birth process (includes intrapartum loss) regardless of route of delivery (Committee on Practice Bulletins-Obstetrics, 2017).
Small for gestational age (singleton/twins) | On the day of delivery.
  Small for gestational age was defined as a birth weight below the 10th percentile (de Onis and Habicht, 1996).
Large for gestational age (singleton/twins) | On the day of delivery.
  Large for gestational age was defined as a birth weight above the 90th percentile.
Birth weight | On the day of delivery.
  In grams; of singletons and twins.
Congenital anomalies | Within 28 days of birth.
  Structural or functional disorders that occur during intra-uterine life and can be identified prenatally, at birth, or later in life. Congenital anomalies can be caused by single gene defects, chromosomal disorders, multifactorial inheritance, environmental teratogens, and micronutrient deficiencies. The time of identification should be reported.
NICU admission | Within 28 days of birth.
  Counting number of babies admited to neonatal intensive care unit.
Reason for NICU admission | Within 28 days of birth.
  Respiratory distress, intraventricular hemorrhagea, necrotizing enterocolitis, or sepsis.
Neonatal mortality rate | Within 28 days of birth.
  Death of a live-born baby within 28 days of birth. This can be divided into early neonatal mortality, if death occurs in the first seven days after birth, and late neonatal if death occurs between eight and 28 days after delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Lan TN Vuong, Assoc. Prof., Principal Investigator — University of Medicine and Pharmacy at Ho Chi Minh City
Locations (2):
- Vietnam (2):
  - My Duc Hospital, Ho Chi Minh City, Ho Chi Minh City
  - My Duc Phu Nhuan Hospital, Ho Chi Minh City, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] ACOG Committee on Obstetric Practice. ACOG practice bulletin. Diagnosis and management of preeclampsia and eclampsia. Number 33, January 2002. American College of Obstetricians and Gynecologists. Int J Gynaecol Obstet. 2002 Apr;77(1):67-75. PMID 12094777
- [Background] Aleyasin A, Aghahosseini M, Safdarian L, Noorzadeh M, Fallahi P, Rezaeian Z, Hoseinimosa S. Can letrozole plus HMG protocol improve pregnancy outcomes in frozen-thawed embryo transfer? An RCT. Int J Reprod Biomed. 2017 Feb;15(2):83-86. PMID 28462399
- [Background] Aslih N, Dorzia D, Atzmon Y, Estrada D, Ellenbogen A, Bilgory A, Shalom-Paz E. Ovulatory-Based FET Cycles May Achieve Higher Pregnancy Rates in the General Population and among Anovulatory Women. J Clin Med. 2021 Feb 11;10(4):703. doi: 10.3390/jcm10040703. PMID 33670133
- [Background] Atkinson M, Crittenden J, Smith H, Sjoblom C. Retrospective cohort study on preparation regimens for frozen embryo transfer. Reprod Fertil. 2021 Nov 23;2(4):308-316. doi: 10.1530/RAF-21-0044. eCollection 2021 Dec. PMID 35118408
- [Background] Bocca-Tjeertes IF, Kerstjens JM, Reijneveld SA, Veldman K, Bos AF, de Winter AF. Growth patterns of large for gestational age children up to age 4 years. Pediatrics. 2014 Mar;133(3):e643-9. doi: 10.1542/peds.2013-0985. Epub 2014 Feb 24. PMID 24567020
- [Background] Braakhekke M, Kamphuis EI, Dancet EA, Mol F, van der Veen F, Mol BW. Ongoing pregnancy qualifies best as the primary outcome measure of choice in trials in reproductive medicine: an opinion paper. Fertil Steril. 2014 May;101(5):1203-4. doi: 10.1016/j.fertnstert.2014.03.047. PMID 24786739
- [Background] Casper RF, Mitwally MF. Use of the aromatase inhibitor letrozole for ovulation induction in women with polycystic ovarian syndrome. Clin Obstet Gynecol. 2011 Dec;54(4):685-95. doi: 10.1097/GRF.0b013e3182353d0f. PMID 22031258
- [Background] Chung TW, Park MJ, Kim HS, Choi HJ, Ha KT. Integrin alphaVbeta3 and alphaVbeta5 are required for leukemia inhibitory factor-mediated the adhesion of trophoblast cells to the endometrial cells. Biochem Biophys Res Commun. 2016 Jan 22;469(4):936-40. doi: 10.1016/j.bbrc.2015.12.103. Epub 2015 Dec 24. PMID 26723254
- [Background] Committee on Practice Bulletins-Obstetrics. Practice Bulletin No. 183: Postpartum Hemorrhage. Obstet Gynecol. 2017 Oct;130(4):e168-e186. doi: 10.1097/AOG.0000000000002351. PMID 28937571
- [Background] Donderwinkel PF, Schoot DC, Pache TD, de Jong FH, Hop WC, Fauser BC. Luteal function following ovulation induction in polycystic ovary syndrome patients using exogenous gonadotrophins in combination with a gonadotrophin-releasing hormone agonist. Hum Reprod. 1993 Dec;8(12):2027-32. doi: 10.1093/oxfordjournals.humrep.a137976. PMID 8150898
- [Background] Duffy JMN, Bhattacharya S, Bhattacharya S, Bofill M, Collura B, Curtis C, Evers JLH, Giudice LC, Farquharson RG, Franik S, Hickey M, Hull ML, Jordan V, Khalaf Y, Legro RS, Lensen S, Mavrelos D, Mol BW, Niederberger C, Ng EHY, Puscasiu L, Repping S, Sarris I, Showell M, Strandell A, Vail A, van Wely M, Vercoe M, Vuong NL, Wang AY, Wang R, Wilkinson J, Youssef MA, Farquhar CM; Core Outcome Measure for Infertility Trials (COMMIT) initiative. Standardizing definitions and reporting guidelines for the infertility core outcome set: an international consensus development study. Fertil Steril. 2021 Jan;115(1):201-212. doi: 10.1016/j.fertnstert.2020.11.013. Epub 2020 Nov 30. PMID 33272619
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S19-S40. doi: 10.2337/dc23-S002. PMID 36507649
- [Background] ESHRE Working Group on Recurrent Implantation Failure; Cimadomo D, de Los Santos MJ, Griesinger G, Lainas G, Le Clef N, McLernon DJ, Montjean D, Toth B, Vermeulen N, Macklon N. ESHRE good practice recommendations on recurrent implantation failure. Hum Reprod Open. 2023 Jun 15;2023(3):hoad023. doi: 10.1093/hropen/hoad023. eCollection 2023. PMID 37332387
- [Background] Franik S, Eltrop SM, Kremer JA, Kiesel L, Farquhar C. Aromatase inhibitors (letrozole) for subfertile women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2018 May 24;5(5):CD010287. doi: 10.1002/14651858.CD010287.pub3. PMID 29797697
- [Background] Ganesh A, Chauhan N, Das S, Chakravarty B, Chaudhury K. Endometrial receptivity markers in infertile women stimulated with letrozole compared with clomiphene citrate and natural cycles. Syst Biol Reprod Med. 2014 Apr;60(2):105-11. doi: 10.3109/19396368.2013.862316. Epub 2013 Dec 5. PMID 24304327
- [Background] Godiwala P, Makhijani R, Bartolucci A, Grow D, Nulsen J, Benadiva C, Grady J, Engmann L. Pregnancy outcomes after frozen-thawed embryo transfer using letrozole ovulation induction, natural, or programmed cycles. Fertil Steril. 2022 Oct;118(4):690-698. doi: 10.1016/j.fertnstert.2022.06.013. Epub 2022 Jul 19. PMID 35863997
- [Background] Haouzi D, Assou S, Mahmoud K, Tondeur S, Reme T, Hedon B, De Vos J, Hamamah S. Gene expression profile of human endometrial receptivity: comparison between natural and stimulated cycles for the same patients. Hum Reprod. 2009 Jun;24(6):1436-45. doi: 10.1093/humrep/dep039. Epub 2009 Feb 26. PMID 19246470
- [Background] Harmsen MJ, Van den Bosch T, de Leeuw RA, Dueholm M, Exacoustos C, Valentin L, Hehenkamp WJK, Groenman F, De Bruyn C, Rasmussen C, Lazzeri L, Jokubkiene L, Jurkovic D, Naftalin J, Tellum T, Bourne T, Timmerman D, Huirne JAF. Consensus on revised definitions of Morphological Uterus Sonographic Assessment (MUSA) features of adenomyosis: results of modified Delphi procedure. Ultrasound Obstet Gynecol. 2022 Jul;60(1):118-131. doi: 10.1002/uog.24786. PMID 34587658
- [Background] Healey S, Tan SL, Tulandi T, Biljan MM. Effects of letrozole on superovulation with gonadotropins in women undergoing intrauterine insemination. Fertil Steril. 2003 Dec;80(6):1325-9. doi: 10.1016/j.fertnstert.2003.03.001. PMID 14667860
- [Background] Hecher K, Diehl W. Chapter 13 - Multiple pregnancies. In Wladimiroff JW, Eik-Nes SH, editors. Ultrasound Obstet Gynaecol 2009. p. 247-258. Elsevier: Edinburgh. Available from: https://www.sciencedirect.com/science/article/pii/B9780444518293000131.
- [Background] Herskovits AZ, Chen Y, Latifi N, Ta RM, Kriegel G. False-Negative Urine Human Chorionic Gonadotropin Testing in the Clinical Laboratory. Lab Med. 2020 Jan 2;51(1):86-93. doi: 10.1093/labmed/lmz039. PMID 31245816
- [Background] Hosseini-Najarkolaei A, Moini A, Kashani L, Farid Mojtahedi M, Hosseini-Najarkolaee E, Salehi E. The effect of letrozole versus artificial hormonal endometrial preparation on pregnancy outcome after frozen-thawed embryos transfer cycles: a randomized clinical trial. Reprod Biol Endocrinol. 2020 Nov 20;18(1):115. doi: 10.1186/s12958-020-00675-z. PMID 33218350
- [Background] Hu YJ, Chen YZ, Zhu YM, Huang HF. Letrozole stimulation in endometrial preparation for cryopreserved-thawed embryo transfer in women with polycystic ovarian syndrome: a pilot study. Clin Endocrinol (Oxf). 2014 Feb;80(2):283-9. doi: 10.1111/cen.12280. Epub 2013 Jul 24. PMID 23808904
- [Background] Khadem Ghaebi N, Mahmoudiniya M, Najaf Najafi M, Zohdi E, Attaran M. Comparison of letrozole with gonadotropin-releasing hormone agonist in frozen embryo transfer after recurrent implantation failure: An RCT. Int J Reprod Biomed. 2020 Feb 27;18(2):105-112. doi: 10.18502/ijrm.v18i2.6417. eCollection 2020 Feb. PMID 32259004
- [Background] Li SJ, Zhang YJ, Chai XS, Nie MF, Zhou YY, Chen JL, Tao GS. Letrozole ovulation induction: an effective option in endometrial preparation for frozen-thawed embryo transfer. Arch Gynecol Obstet. 2014 Mar;289(3):687-93. doi: 10.1007/s00404-013-3044-0. Epub 2013 Oct 10. PMID 24121690
- [Background] Lin J, Wang N, Huang J, Cai R, Fan Y, Kuang Y, Wang Y. Pregnancy And Neonatal Outcomes Of hMG Stimulation With Or Without Letrozole In Endometrial Preparation For Frozen-Thawed Embryo Transfer In Ovulatory Women: A Large Retrospective Cohort Study. Drug Des Devel Ther. 2019 Nov 14;13:3867-3877. doi: 10.2147/DDDT.S212235. eCollection 2019. PMID 31814708
- [Background] Lou L, Xu Y, Lv M, Yu J, Xiao Q, Chen P, Bai M, Zhang Z. Comparison of different endometrial preparation protocols on frozen embryo transfer pregnancy outcome in patients with normal ovulation. Reprod Biomed Online. 2022 Dec;45(6):1182-1187. doi: 10.1016/j.rbmo.2022.06.026. Epub 2022 Jul 4. PMID 36085270
- [Background] Macrosomia: ACOG Practice Bulletin, Number 216. Obstet Gynecol. 2020 Jan;135(1):e18-e35. doi: 10.1097/AOG.0000000000003606. PMID 31856124
- [Background] Miller PB, Parnell BA, Bushnell G, Tallman N, Forstein DA, Higdon HL 3rd, Kitawaki J, Lessey BA. Endometrial receptivity defects during IVF cycles with and without letrozole. Hum Reprod. 2012 Mar;27(3):881-8. doi: 10.1093/humrep/der452. Epub 2012 Jan 13. PMID 22246449
- [Background] Montville CP, Khabbaz M, Aubuchon M, Williams DB, Thomas MA. Luteal support with intravaginal progesterone increases clinical pregnancy rates in women with polycystic ovary syndrome using letrozole for ovulation induction. Fertil Steril. 2010 Jul;94(2):678-83. doi: 10.1016/j.fertnstert.2009.03.088. Epub 2009 Jun 9. PMID 19515366
- [Background] Munro MG, Critchley HO, Broder MS, Fraser IS; FIGO Working Group on Menstrual Disorders. FIGO classification system (PALM-COEIN) for causes of abnormal uterine bleeding in nongravid women of reproductive age. Int J Gynaecol Obstet. 2011 Apr;113(1):3-13. doi: 10.1016/j.ijgo.2010.11.011. Epub 2011 Feb 22. PMID 21345435
- [Background] Niu Y, Zhao D, Wang Y, Suo L, Zou J, Wei D. Ovulation induction regimens are associated with a higher rate of livebirth after frozen single-blastocyst transfer among women with polycystic ovary syndrome. Front Endocrinol (Lausanne). 2022 Aug 15;13:987813. doi: 10.3389/fendo.2022.987813. eCollection 2022. PMID 36046783
- [Background] de Onis M, Habicht JP. Anthropometric reference data for international use: recommendations from a World Health Organization Expert Committee. Am J Clin Nutr. 1996 Oct;64(4):650-8. doi: 10.1093/ajcn/64.4.650. PMID 8839517
- [Background] Oxford Textbook of Obstetrics and Gynaecology 2020; Oxford University Press Available from: https://academic.oup.com/book/29679.
- [Background] Pathirana J, Munoz FM, Abbing-Karahagopian V, Bhat N, Harris T, Kapoor A, Keene DL, Mangili A, Padula MA, Pande SL, Pool V, Pourmalek F, Varricchio F, Kochhar S, Cutland CL; Brighton Collaboration Neonatal Death Working Group. Neonatal death: Case definition & guidelines for data collection, analysis, and presentation of immunization safety data. Vaccine. 2016 Dec 1;34(49):6027-6037. doi: 10.1016/j.vaccine.2016.03.040. Epub 2016 Jul 19. PMID 27449077
- [Background] Pfeifer SM, Attaran M, Goldstein J, Lindheim SR, Petrozza JC, Rackow BW, Siegelman E, Troiano R, Winter T, Zuckerman A, Ramaiah SD. ASRM mullerian anomalies classification 2021. Fertil Steril. 2021 Nov;116(5):1238-1252. doi: 10.1016/j.fertnstert.2021.09.025. PMID 34756327
- [Background] Rezk M, Hamza H, El-Shamy ES. Luteal support with vaginal dydrogesterone increases pregnancy rate in patients with clomifene resistant polycystic ovary syndrome receiving letrozole for ovulation induction. Gynecol Endocrinol. 2019 Mar;35(3):217-219. doi: 10.1080/09513590.2018.1512571. Epub 2018 Oct 16. PMID 30324834
- [Background] Royal College of Obstetricians and Gynaecologists. Antepartum Haemorrhage (Green-top Guideline No. 63). 2011; Available from: https://www.rcog.org.uk/guidance/browse-all-guidance/green-top-guidelines/antepartum-haemorrhage-green-top-guideline-no-63/.
- [Background] Samsami A, Ghasmpour L, Davoodi S, Moradi Alamdarloo S, Rahmati J, Karimian A, Homayoon H. Frozen embryo transfer: Endometrial preparation by letrozole versus hormone replacement cycle: A randomized clinical trial. Int J Reprod Biomed. 2019 Dec 30;17(12):915-922. doi: 10.18502/ijrm.v17i12.5793. eCollection 2019 Dec. PMID 31970313
- [Background] Simon C, Cano F, Valbuena D, Remohi J, Pellicer A. Clinical evidence for a detrimental effect on uterine receptivity of high serum oestradiol concentrations in high and normal responder patients. Hum Reprod. 1995 Sep;10(9):2432-7. doi: 10.1093/oxfordjournals.humrep.a136313. PMID 8530680
- [Background] Sotiriadis A, Papatheodorou S, Makrydimas G. Threatened miscarriage: evaluation and management. BMJ. 2004 Jul 17;329(7458):152-5. doi: 10.1136/bmj.329.7458.152. No abstract available. PMID 15258071
- [Background] Teede HJ, Misso ML, Costello MF, Dokras A, Laven J, Moran L, Piltonen T, Norman RJ; International PCOS Network. Recommendations from the international evidence-based guideline for the assessment and management of polycystic ovary syndrome. Fertil Steril. 2018 Aug;110(3):364-379. doi: 10.1016/j.fertnstert.2018.05.004. Epub 2018 Jul 19. PMID 30033227
- [Background] Teede HJ, Tay CT, Laven JJE, Dokras A, Moran LJ, Piltonen TT, Costello MF, Boivin J, Redman LM, Boyle JA, Norman RJ, Mousa A, Joham AE. Recommendations From the 2023 International Evidence-based Guideline for the Assessment and Management of Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2023 Sep 18;108(10):2447-2469. doi: 10.1210/clinem/dgad463. PMID 37580314
- [Background] Wang X, Chen C, Wang L, Chen D, Guang W, French J. Conception, early pregnancy loss, and time to clinical pregnancy: a population-based prospective study. Fertil Steril. 2003 Mar;79(3):577-84. doi: 10.1016/s0015-0282(02)04694-0. PMID 12620443
- [Background] Webster K, Fishburn S, Maresh M, Findlay SC, Chappell LC; Guideline Committee. Diagnosis and management of hypertension in pregnancy: summary of updated NICE guidance. BMJ. 2019 Sep 9;366:l5119. doi: 10.1136/bmj.l5119. No abstract available. PMID 31501137
- [Background] Zegers-Hochschild F, Adamson GD, Dyer S, Racowsky C, de Mouzon J, Sokol R, Rienzi L, Sunde A, Schmidt L, Cooke ID, Simpson JL, van der Poel S. The International Glossary on Infertility and Fertility Care, 2017. Hum Reprod. 2017 Sep 1;32(9):1786-1801. doi: 10.1093/humrep/dex234. PMID 29117321
- [Background] Zeng MF, Zhou X, Duan JL. Stimulated cycle versus artificial cycle for frozen embryo transfer in patients with polycystic ovary syndrome: a Meta-analysis. Gynecol Endocrinol. 2021 Apr;37(4):294-299. doi: 10.1080/09513590.2020.1867976. Epub 2021 Jan 10. PMID 33426930
- [Background] Zhang J, Li Z, Sun L, Guan Y, Du M. Comparison of Pregnancy and Neonatal Outcomes of Single Frozen Blastocyst Transfer Between Letrozole-Induction and HRT Cycles in Patients With Abnormal Ovulation. Front Endocrinol (Lausanne). 2021 Apr 16;12:664072. doi: 10.3389/fendo.2021.664072. eCollection 2021. PMID 33935972
- [Background] Zhang J, Wang L, Li C, Zhang H, Li R, Li M. Letrozole promotes the expression of integrin alphavbeta3 and HOXA10 in endometrium of endometriosis. Syst Biol Reprod Med. 2022 Apr;68(2):121-128. doi: 10.1080/19396368.2021.2013577. Epub 2021 Dec 28. PMID 34962452
- [Background] Zhang J, Wei M, Bian X, Wu L, Zhang S, Mao X, Wang B. Letrozole-induced frozen embryo transfer cycles are associated with a lower risk of hypertensive disorders of pregnancy among women with polycystic ovary syndrome. Am J Obstet Gynecol. 2021 Jul;225(1):59.e1-59.e9. doi: 10.1016/j.ajog.2021.01.024. Epub 2021 Jan 30. PMID 33529574
- [Background] Zhang W, Liu Z, Zhang J, Ren B, Liu M, Li J, Zhang W, Guan Y. Comparison of Perinatal Outcomes of Letrozole-Induced Ovulation and Hormone Replacement Therapy Protocols in Patients With Abnormal Ovulation Undergoing Frozen-Thawed Embryo Transfer: A Propensity Score Matching Analysis. Front Endocrinol (Lausanne). 2022 Mar 16;13:837731. doi: 10.3389/fendo.2022.837731. eCollection 2022. PMID 35370976
- [Background] Zhang Y, Fu X, Gao S, Gao S, Gao S, Ma J, Chen ZJ. Preparation of the endometrium for frozen embryo transfer: an update on clinical practices. Reprod Biol Endocrinol. 2023 Jun 8;21(1):52. doi: 10.1186/s12958-023-01106-5. PMID 37291605
- [Background] Zhang Y, Wu L, Li TC, Wang CC, Zhang T, Chung JPW. Systematic review update and meta-analysis of randomized and non-randomized controlled trials of ovarian stimulation versus artificial cycle for endometrial preparation prior to frozen embryo transfer in women with polycystic ovary syndrome. Reprod Biol Endocrinol. 2022 Apr 2;20(1):62. doi: 10.1186/s12958-022-00931-4. PMID 35366912